CLINICAL TRIAL: NCT00897884
Title: Clinical and Biologic Effects of Metformin in Early Stage Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mount Sinai Hospital, Canada (Other)
Collaborators: Princess Margaret Hospital, Canada (Other)
Responsible Party: Dr. Pamela Goodwin, Mount Sinai Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: METFORMIN
Record Dates: First submitted 2009-05-08; First posted 2009-05-12 (Estimated); Last update posted 2012-01-19 (Estimated); Status verified 2012-01

CONDITIONS: Breast Cancer
Keywords: breast cancer; metformin; breast surgery
MeSH Terms: conditions — Breast Neoplasms | interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Metformin (Experimental): Patients will take metformin three times a day for two to three weeks prior surgery.
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Metformin — 500 mg tablet, taken 3 times a day for 2-3 weeks

SUMMARY:
The study will be testing metformin in patients with breast cancer who are about to undergo surgery. Patients will take metformin 3 times daily for about 2-3 weeks prior to their surgery date. It is hypothesized that metformin will reduce cell proliferation rates in tumour tissue.

ELIGIBILITY:
Inclusion Criteria:

1. invasive T1-4 (if T1, ≥ 1cm), NX operable breast cancer confirmed on core biopsy
2. < 70 years of age
3. breast surgery scheduled at least 2 weeks after study entry at one of the participating institutions (metformin will be started no more than 3 weeks prior to scheduled surgery) for the current breast cancer
4. patient and physician consent

Exclusion Criteria:

1. on metformin for any reason during the preceding 4 weeks
2. recent (within 4 weeks) antiestrogen or estrogen therapy
3. prior or concurrent systemic neoadjuvant BC therapy of any type (chemotherapy, hormone therapy, biologic therapy)
4. known diabetes or baseline fasting glucose > or = 7.0 mmol/L (specific treatment is required)
5. current or recent (within 4 weeks) use of drugs that may influence insulin or insulin sensitivity including oral corticosteroids, insulin sensitizers, exogenous insulin or oral hypoglycemic agents
6. serum creatinine above upper limit of normal for the institution
7. history of lactic or other metabolic acidosis
8. consumption of > 3 alcoholic beverages per day (on average)
9. AST > 1.5 times upper limit of normal for the institution
10. known hypersensitivity or allergy to metformin
11. current or past congestive heart failure
12. coagulopathy (including use of anti-coagulants) precluding biopsy
13. pregnancy or lactation within 3 months.
14. Serious psychiatric illness

    * Note: Women with childbearing potential will be required to use an effective form of birth control (condom or other barrier method, tubal ligation or vasectomy - oral contraceptives are contra-indicated in breast cancer) and to have a negative pregnancy test prior to starting metformin.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2008-10; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
To determine if taking metformin prior to surgery can reduce cell proliferation rates in tumour tissue. To be determined by tumour specimen analysis using pre- and post-operative biopsy sample. | two to three weeks

CONTACTS AND LOCATIONS:
Overall Officials: Pamela J Goodwin, MD, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (2):
- Canada (2):
  - Mount Sinai Hospital, Toronto, Ontario
  - Princess Margaret Hospital, Toronto, Ontario

REFERENCES:
- [Derived] Dowling RJ, Niraula S, Chang MC, Done SJ, Ennis M, McCready DR, Leong WL, Escallon JM, Reedijk M, Goodwin PJ, Stambolic V. Changes in insulin receptor signaling underlie neoadjuvant metformin administration in breast cancer: a prospective window of opportunity neoadjuvant study. Breast Cancer Res. 2015 Mar 3;17(1):32. doi: 10.1186/s13058-015-0540-0. PMID 25849721